CLINICAL TRIAL: NCT00382733
Title: Oral Topotecan, Utilization for a Metronomic Dosing Schedule to Treat Recurrent or Persistent Solid Tumors
Brief Title: Oral Topotecan to Treat Recurrent or Persistent Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ATDTROC0501
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Tumors
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral Topotecan — Topotecan will be received in one of the five dose levels:0.25mg/day,0.5mg/day, 0.75mg/day, 1.0mg/day, and 1.25mg/day.
  Other Names: Hycamtin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of oral topotecan and how well the chemotherapy is tolerated (any side effects) when it is given in different dose levels. The study will also collect information on how the medication is being broken down and absorbed in the body and how quality of life is affected during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Male or female patients.
* Patient is at least 18 years of age with recurrent or persistent solid tumors.
* Patient has adequate hematologic function (absolute neutrophil count [ANC] >= 1500/mL and platelets >= 100,000/mL), adequate renal function (serum creatinine < 2.0 mg/dL; calculated creatinine clearance > 40 mL/min), and adequate hepatic function (serum bilirubin <= 1.5 mg/dL and transaminases <= 3 times the upper limit of normal [3 x ULN]).
* Patient has Eastern Oncology Cooperative Group (ECOG) performance status of <= 2.
* Patient has a life expectancy of at least 3 months at time of enrollment.
* Patient has no medical problems, unrelated to the malignancy, of sufficient severity which would limit full compliance with the study or which would expose him/her to undue risks.
* Patient has received no more than 2 prior treatment regimens prior to enrollment including chemotherapy, hormonal therapy, biologic therapy, and immunotherapy.
* Patient has a negative serum or urine pregnancy test within 7 days prior to starting therapy (if a female of childbearing potential).

Exclusion Criteria:

* Patient is a pregnant or lactating woman. Women of childbearing potential with either a positive or no pregnant test (serum or urine) at baseline. Women of childbearing potential not using a reliable and appropriate contraceptive method will be excluded. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.) Patients must agree to continue contraception for 30 days from the date of the last study drug administration.
* Patient has serious, uncontrolled, concurrent infection(s).
* Patient has received whole pelvic or extended field radiation therapy within 4 weeks of enrollment. Patients who have not fully recovered or whose acute toxicity related to prior radiotherapy has not returned to baseline are ineligible.
* Patient has received myelosuppressive chemotherapy within the last 4 weeks or has not recovered from the myelosuppressive effects of recent chemotherapy.
* Patient has received another investigational agent within 4 weeks prior to study enrollment.
* Patient has known hypersensitivity to topoisomerase I inhibitors.
* Patient is unable to swallow a capsule or has a disease known to affect drug absorption, such as short gut syndrome or active radiation enteritis.
* Patient has received drugs known to alter absorption such as antacids, proton pump blockers (eg, omeprazole), or H2 receptor antagonists (eg, cimetidine). A washout period of one week (7 days) is required prior to initiating study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd D. Tillmanns, M.D., Principal Investigator — West Clinic
Locations (1):
- The West Clinic, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to enrollment at one community oncology clinic from November 2006 to May 2009.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening period that could last up to 4 weeks during which pre-study assessments were completed. During the dose finding portion of the study, subjects were assigned to a Dose Level during enrollment. Once the MTD was determined, additional subjects were treated at the MTD.
Groups:
- Oral Topotecan 0.25 mg Daily: All subjects in this group were assigned to receive metronomic oral topotecan 0.25 mg daily (Dose Level 1).
- Oral Topotecan 0.50 mg Daily: All subjects in this group were assigned to receive metronomic oral topotecan 0.50 mg daily (Dose Level 2).
- Oral Topotecan 0.75 mg Daily: All subjects in this group were assigned to receive metronomic oral topotecan 0.75 mg daily (Dose Level 3).
- Oral Topotecan 1.0 mg Daily: All subjects in this group were assigned to receive metronomic oral topotecan 1.0 mg daily (Dose Level 4).
- Oral Topotecan 1.25 mg Daily: All subjects in this group were assigned to receive metronomic oral topotecan 1.25 mg daily (Dose Level 5).
Period: Overall Study
Arm/Group | Oral Topotecan 0.25 mg Daily | Oral Topotecan 0.50 mg Daily | Oral Topotecan 0.75 mg Daily | Oral Topotecan 1.0 mg Daily | Oral Topotecan 1.25 mg Daily
Started | 3 | 4 | 3 | 14 | 2
Completed | 3 | 3 (1 subject withdrew consent before completing Cycle 1 - that subject was replaced) | 3 | 14 | 2
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metronomic Oral Topotecan: All subjects received metronomic oral topotecan daily at the assigned dose level.
Arm/Group | Metronomic Oral Topotecan
Number analyzed (Participants) | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Single Agent Metronomic Oral Topotecan
Description: The MTD of metronomic oral topotecan was determined using a standard 3+3 dose escalation cohort design. The total sample and the number of subjects who receive each dose in this design depends on the frequency of dose limiting toxicities (DLTs)at each dose level. If 0 out of 3 subjects experience a DLT at a given dose level, 3 subjects will be enrolled at the next higher dose level. If greater than or equal to 2 subjects experience a DLT at a given dose level, dose escalation will be stopped. If 1 out of 3 subjects experience a DLT at a given dose level, 3 subjects are enrolled at the same dose level.
Time Frame: MTD was assessed during the first cycle of treatment (days 1-28).
Population: DLT information was available for 3 subjects who received a topotecan dose of 0.25 mg/day, 3 subjects who received a topotecan dose of 0.50 mg/day, 3 subjects who received a topotecan dose of 0.75 mg/day, 3 subjects who received a topotecan dose of 1.0 mg/day, and 2 subjects who received a topotecan dose of 1.25 mg/day.
Measure: Number; unit: mg/day
Arm/Group | Metronomic Oral Topotecan
Number analyzed (Participants) | 14
mg/day | 1.0

2. Secondary Outcome: Dose Limiting Toxicities (DLT)
Description: DLTs were assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. This measure reports the number of subjects who experienced DLT at each dose level during the dose finding portion of the study.
Time Frame: DLTs were assessed during the first cycle of treatment (days 1-28).
Population: Number of participants analyzed refers to those for whom DLT information was available during the dose finding portion of the study.
Measure: Number; unit: participants
Arm/Group | Oral Topotecan 0.25 mg Daily | Oral Topotecan 0.50 mg Daily | Oral Topotecan 0.75 mg Daily | Oral Topotecan 1.0 mg Daily | Oral Topotecan 1.25 mg Daily
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
participants | 0 | 0 | 0 | 0 | 2

3. Secondary Outcome: Best Overall Response
Description: Best overall response is defined as the best response across all time points. Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of disease progression. Response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Best overall response was assessed after every 8 weeks of treatment and at the end of treatment or time of disease progression, up to 1 year.
Population: All enrolled subjects were analyzed for this outcome.
Measure: Number; unit: participants
Arm/Group | Oral Topotecan 0.25 mg Daily | Oral Topotecan 0.50 mg Daily | Oral Topotecan 0.75 mg Daily | Oral Topotecan 1.0 mg Daily | Oral Topotecan 1.25 mg Daily
Number analyzed (Participants) | 3 | 4 | 3 | 14 | 2
participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1 | 0
  Stable Disease | 2 | 1 | 2 | 4 | 0
  Progressive Disease | 0 | 1 | 1 | 2 | 0
  Not Evaluable | 1 | 2 | 0 | 7 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected on day 1 of treatment until one month after the end of study treatment.
Description: Subjects were systematically assessed for adverse events on day 1 of each cycle by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Oral Topotecan 0.25 mg Daily | Oral Topotecan 0.50 mg Daily | Oral Topotecan 0.75 mg Daily | Oral Topotecan 1.0 mg Daily | Oral Topotecan 1.25 mg Daily
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 0/3 | 7/14 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 13/14 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Topotecan 0.25 mg Daily (N=3) | Oral Topotecan 0.50 mg Daily (N=4) | Oral Topotecan 0.75 mg Daily (N=3) | Oral Topotecan 1.0 mg Daily (N=14) | Oral Topotecan 1.25 mg Daily (N=2)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Topotecan 0.25 mg Daily (N=3) | Oral Topotecan 0.50 mg Daily (N=4) | Oral Topotecan 0.75 mg Daily (N=3) | Oral Topotecan 1.0 mg Daily (N=14) | Oral Topotecan 1.25 mg Daily (N=2)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Eye hemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 6 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 7 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 1 | 7 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral edema (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Waist circumference increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less